CLINICAL TRIAL: NCT07269951
Title: Assessment of Bone Thickness in the Infrazygomatic Crest and Proper Insertion Angle for Miniscrew Positioning: A Retrospective CBCT Study
Brief Title: The Bone Thickness of Infrazygomatic Crest Was Measured on CBCTs
Acronym: IZC
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fady Hussein, Professor, Cairo University
Other Study IDs: 31-3-22
Record Dates: First submitted 2025-08-23; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Miniscrew Placement
Keywords: miniscrew; TAD; infrazygomatic crest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 95 patients were randomly chosen constituting both males and females: Following the inclusion and exclusion criteria, 95 patients were randomly chosen constituting both males and females with an age range of 20-35 years old (58 females and 37 males). CBCTs were acquired in the same manner, using an i-CAT scanner with 110 kVp, 60 mA, 0.3-mm voxel size, a scan time of 18 seconds, and a field of view of 17x 23 cm. CBCT measurements were analyzed using Invivo 6 (Anatomage, Inc., Santa Clara, Calif). These tomographic images were reoriented so that the natural head position coincided with the true horizontal plane in an attempt to reduce possible errors in head positioning during image acquisition.

SUMMARY:
This study will be done on 95 patients with CBCTs retrospectively, to evaluate the bone depth of infrazygomatic crest region for selecting suitable size of miniscrews and proper insertion angle clinical guide in the infrazygomatic crest without injuring the mesiobuccal root of the maxillary first molar.

DETAILED DESCRIPTION:
CBCTs of 95 patients were collected retrospectively from archives of Faculty of Dentistry, Cairo University, that were requested for different dental purposes. The thickness of the IZC was measured above mesio-buccal root of upper 6 (U6MB), above disto-buccal root of upper 6 (U6DB) and contact point between upper 6 and 7 roots (U6-7). The distance from point of entry of miniscrew to the occlusal plane, that saves roots from injury, was measured. Then, the angle of miniscrew insertion in relation to the occlusal plane was measured at maximum thickness available together with point of entry in relation to the occlusal plane. The IZC thickness of right and left sides of each patient was compared, also compared in males and females. Kruskal-Wallis test, Paired Wilcoxon signed rank test & Spearman correlation were used to analyze results

ELIGIBILITY:
Inclusion Criteria:

* Patients having full permanent dentition
* all cases were indicated for CBCT for their orthodontic treatment
* Patients with sound dentition

Exclusion Criteria:

* craniofacial anomalies and facial asymmetries
* Unclear CBCT
* mixed dentition
* Patients with systemic bone disorders

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be done on 100 CBCTs of 95 patients; 58 females and 37 males retrospectively to evaluate the bone depth of infrazygomatic crest region for selecting suitable size of miniscrews and proper insertion angle clinical guide in the infrazygomatic crest without injuring the mesiobuccal root of the maxillary first molar.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
measure bone thickness of infrazygomatic crest | from enrollment to the end of taking measurements at 8 weeks
  the bone thickness will be measured on CBCT from coronal slice at 3 points : above mesio-buccal root of upper first molar, above disto-buccal root of upper first molar and between upper first and second molars contact points

SECONDARY OUTCOMES:
proper angulation of miniscrew insertion | from enrollment to the end of taking measurements at 8 weeks
  a clinical guide to clinicians was done to guide the clinician the proper angulation of long axis of miniscrew and occlusal plane
check asymmetry of right and left sides per patient | from enrollment to the end of taking measurements at 8 weeks
  the right and left bone thickness was measured to detect any asymmetry between both sides

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
mean age of the patients mean thickness of infrazygomatic crest
Time Frame: start date for IPD sharing : 1 December, 2025 start date for IPD sharing : 1 December, 2026
Access Criteria: anyone will be able to access the IPD and supporting information, they will be able to access study protocol, they will be able to access it by sending Email to fady.fahim@gmail.com

REFERENCES:
- [Result] Husseini B, Younes R, Baumgaertel S, El Wak T, El Osta N, Bassil-Nassif N, Bouserhal J. Assessment of infrazygomatic crest dimensions in different vertical facial growth types for miniscrew insertion: A cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2022 Dec;162(6):917-926. doi: 10.1016/j.ajodo.2021.07.029. Epub 2022 Sep 13. PMID 36109268
- [Result] Lima A Jr, Domingos RG, Cunha Ribeiro AN, Rino Neto J, de Paiva JB. Safe sites for orthodontic miniscrew insertion in the infrazygomatic crest area in different facial types: A tomographic study. Am J Orthod Dentofacial Orthop. 2022 Jan;161(1):37-45. doi: 10.1016/j.ajodo.2020.06.044. Epub 2021 Aug 12. PMID 34391619
- [Result] Hijazi Muwaquet K, Muwaquet Rodriguez S, Ferrer Molina M, Hijazi Alsadi T. Optimizing Infrazygomatic Miniscrew Insertion Parameters: Systematic Review and Meta-Regression Analysis of Bone Thickness by Insertion Height, Angulation, and Anatomical Position. J Clin Med. 2025 Jun 5;14(11):4005. doi: 10.3390/jcm14114005. PMID 40507767